CLINICAL TRIAL: NCT06322979
Title: Comparative Evaluation of Premixed Bioceramic Putty Versus MTA as Apical Plugs in Nonvital Immature Anterior Teeth: A Clinical Randomized Controlled Trial
Brief Title: Premixed Bioceramic Putty as an Apical Plug in Immature Anterior Permanent Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shaimaa Shaban Mohamed El-desouky, Lecturer of Pediatric dentistry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: # R-PED-11-23-3074
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Periapical Periodontitis
Keywords: immature teeth; apexification; apical plug
MeSH Terms: conditions — Periapical Periodontitis | interventions — mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MTA group (Active Comparator): After the endodontic procedure, MTA will be placed into the apical 4 mm of the root canals. then a moist cotton pellet will be placed and the access cavity will be restored with GIC. Next day, GIC and the cotton pellet will be removed the coronal and middle third of the root canal will be filled with gutta-percha. The coronal restoration will be completed with GIC, composite.
  Interventions: Procedure: Mineral trioxide aggregate
- Premixed Bioceramic Putty group (Experimental): After the endodontic procedure, Premixed Bioceramic Putty (Well-Root™ PT) will be placed into the apical 4mm of the canals. After 12 min, the coronal and middle third of the root canal will be filled with gutta-percha. The coronal restoration will be completed with GIC, composite.
  Interventions: Procedure: Premixed Bioceramic Putty

INTERVENTIONS:
Procedure: Mineral trioxide aggregate — Apexification treatment was done with mineral trioxide aggregate
  Arms: MTA group
Procedure: Premixed Bioceramic Putty — Apexification treatment was done with Premixed Bioceramic Putty (Well-Root™ PT)
  Arms: Premixed Bioceramic Putty group

SUMMARY:
Following the randomization procedure, children will be divided into 2 groups (25 immature anterior permanent incisors in each group): Group I will be treated with MTA as apical plug while group II will be treated with Premixed Bioceramic Putty as apical plug. After working length determination, instrumentation, and irrigation of the root canals, apical plug will be done. in MTA Group, MTA will be placed into the apical 4 mm of root canals, then a moist cotton pellet will be placed and the access cavity will be restored with glass-ionomer-based restoration. Next day, glass-ionomer-based restoration and the cotton pellet will be removed, then the coronal restoration will be completed with GIC, composite. In the Premixed Bioceramic Putty group, Well-Root™ PT will be placed into the apical 4 mm of the canals. After 12 min, the coronal and middle third of the root canal will be filled with gutta-percha. The coronal restoration will be completed with GIC, composite.

children will be recalled for clinical and radiographical follow-up after 6 and12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* nonvital immature permanent teeth as a consequence of trauma or dental caries
* nonvital permanent teeth with radiographic evidence of immature root end development
* clinically restorable teeth

Exclusion Criteria:

* immature nonvital permanent teeth presenting with signs/symptoms of internal/external resorption, moderate to severe mobility, periodontal bone loss
* Immature nonvital permanent teeth associated with developmental abnormalities.
* Patients with a history of systemically debilitating diseases
* unrestorable remaining crown structure

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
the clinical success of apexification after using a new apical plug material (Premixed Bioceramic Putty ) compared to the widely used material (MTA) | up to 12 months
  The apexification procedure will be recorded as a clinical success if the tooth fulfils the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility.
the radiographic success of apexification after using a new apical plug material (Premixed Bioceramic Putty ) compared to the widely used material (MTA) | at 6 and12 months follow up
  The apexification procedure will be recorded to be radiographically successful if it demonstrates the following criteria: (1) reduction of apical lesion size (2) Normal periodontal ligament space (2) No furcation pathosis, and (3) No external resorption.
  The apexification procedure will be radiographically unsuccessful if the apical lesion size increases.
  The apexification procedure will be doubtful if the apical lesion size doesn't change

SECONDARY OUTCOMES:
Change in the periapical index (PAI) | at 6 and12 months follow up
  Radio-graphically, the periapical index provides an ordinal scale of 5 scores ranging from ''healthy'' to ''severe periodontitis with exacerbating features''. (1) Normal periapical structures. (2) Small changes in bone structure. (3) Changes in bone structure with some diffuse mineral loss. (4) Periodontitis with well-deﬁned radiolucent area. (5) Severe periodontitis with exacerbating features. (1, 2: healthy and 3, 4, 5: pathological).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698